CLINICAL TRIAL: NCT05571384
Title: High Intensity Body-weight Circuit Training Feasibility and Efficacy for Improving Metabolic Profile, Body Composition, and Health-Related Fitness in Middle Aged Persons With Type 2 Diabetes
Brief Title: High Intensity Body-weight Circuit Training Feasibility and Efficacy for in Middle Aged Persons With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kennesaw State University (Other)
Responsible Party: Principal Investigator, Brian Kliszczewicz, Associate Professor, Kennesaw State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KennesawSU
Record Dates: First submitted 2022-09-23; First posted 2022-10-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Type2diabetes
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high intensity body-weight circuit (HIBC) (Experimental): HIBC Exercise Protocol- circuit repetition and order is as follows: modified squats (10 repetitions), modified rows (5 repetitions), crunches (10), and modified push-ups (5). The exercise sessions will involve repeating a series of repetitions of each movement in sequence, and completing as many sequences as possible in good form in the time allotted for the exercise (initially, 5 minutes). Three sessions per week will be completed at home. After three weeks of training, participants will be asked to add a fourth session each week. Initially, the HIBC sessions will be five minutes long, and the duration of the sessions will increase by one minute each week as tolerated beginning in week four, peaking at 10-minutes per session (warm up not included in this timing) as early as the eighth week of training. Session duration will be capped at 10-minutes.
  Interventions: Behavioral: high intensity body-weight circuit

INTERVENTIONS:
Behavioral: high intensity body-weight circuit — Bodyweight and suspension training equipment (TRX® Fit System) with modified movements. Modified Squats: participants will be instructed to hold the handles of the band with arms extended, participants will then lean back in a standing position and perform a squat within a comfortable range of motion while weight is being distributed to the band. Modified Rows: participants will grab the bands with arms and legs extended. They will find a comfortable angle by which to perform a "row" (pulling the handles to the rib cage) with arms at a 45-degree angle. Modified Push-Ups: perform push-ups on their knees with a flat back and hands underneath their shoulders. They will be instructed to lower their chest towards the ground in a controlled manner and as far as comfort will allow them. Modified Crunches: participants will lay on their back with feet approximately 8-10 inches from their buttocks, and asked to lift their shoulders slightly off the ground.

SUMMARY:
This research study proposes to quantify the efficacy of the novel high intensity body-weight circuit (HIBC) training intervention on metabolic profile, body composition, and health related fitness exercise in middle aged persons with type-2 diabetes (T2DM). This research project is extremely relevant to public health, in that prevalence of T2DM continues to rise on a national and global scale, placing a heavy economic cost on both the healthcare industry and the individual patient in an age-dependent fashion. Results of this study may provide an effective and appealing alternative exercise intervention for cardiometabolic disease management in adults with T2DM, and have significant clinical and public health applications.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosed of type 2 diabetes (T2DM) (within a year) * HbA1c of 6% or higher

  * Non-insulin dependent
  * No medicinal treatment
  * Not currently undergoing a physical activity program in the last six months
  * Received written medical clearance from overseeing physician

Exclusion Criteria:

* Those who have undergone any revascularization procedure

  * Diagnosed with or symptomatic of any renal, pulmonary, or cardiovascular disease (CVD)
  * Diagnosed cognitive dysfunction
  * Current smoker

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
HbA1c change within participant | Pre and post 16-week intervention
  HbA1c (glycosylated Hemoglobin) indicates what the blood glucose environment was like for that past 3-months. This is the average life span of a red blood cell. High levels of blood glucose over a 3 month period lead to high HbA1c and vis versa. HbA1c can change as early as 14 weeks.
Oral Glucose Tolerance Test change within participant | Pre and post 16-week intervention
  Glucose and Insulin response to bolus amount of glucose beverage
Body Composition change within participant | Pre and post 16-week intervention
  Fat mass and lean mass
Estimated VO2max (oxygen consumption), aerobic exercise capacity change within participant | Pre and post 16-week intervention
  sub maximal treadmill endurance test

CONTACTS AND LOCATIONS:
Locations (1):
- Kennesaw State Univeristy, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No